CLINICAL TRIAL: NCT00998920
Title: Randomized, Double-Blind, Rising Multiple Dose Study of S-Equol in Normal Volunteers
Brief Title: Multi-Dose Safety and Pharmacokinetic Study of S-Equol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ausio Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: AUS-CT02
Record Dates: First submitted 2009-10-12; First posted 2009-10-21 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 10mg BID (Experimental): S-equol capsule, oral, single dose
  Interventions: Drug: S-equol
- 20 mg BID (Experimental)
  Interventions: Drug: S-equol
- 40mg BID (Experimental)
  Interventions: Drug: S-equol
- 80 mg BID (Experimental)
  Interventions: Drug: S-equol
- 160 mg BID (Experimental)
  Interventions: Drug: S-equol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-equol — oral, BID, 14 days
  Other Names: AUS-131
  Arms: 10mg BID; 160 mg BID; 20 mg BID; 40mg BID; 80 mg BID
Drug: Placebo — oral, BID, 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating multiple doses of S-equol administered twice daily (BID) for 14 days to healthy male and female subjects and to describe the pharmacokinetic profile of S-equol.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled trial of doses escalated by cohort. Volunteers will be randomized to receive active study drug or placebo twice daily (BID) for 14 days. This study will be staggered in timing with the single rising dose study (Protocol AUS-CT01) being conducted concurrently, such that the lowest dose cohort of this multiple rising dose study may begin after evaluation of safety and pharmacokinetic data from the first 8 subjects randomized to the 10 mg dose cohort of the single rising dose study and safety data from the 8 Subjects randomized in the 20 mg dose cohort of that study.

ELIGIBILITY:
Inclusion Criteria:

* subject is capable of reading, understanding and complying with the protocol and has signed the informed consent document prior to undergoing any study related procedures;
* subject is male or female and is 18 (at the time of consent) to 65 years of age, inclusive (subjects are required to meet the latter age limits by the time of first dosing);
* subject, if female, must be non-lactating, and have a negative serum pregnancy test result during the Pretreatment Period. Women of child-bearing potential must be willing to stay in the clinic from Day -10 until the end of the dosing period to confirm non-pregnant status.
* subject, if female, must be surgically sterile (must be documented); post-menopausal (defined as at least 2 years without menses with screening FSH in expected range) or must be using acceptable methods of non-hormonal contraception (Mirena is acceptable). For this study, estrogen-containing contraceptives are not acceptable. Postmenopausal women must not have had any vaginal spotting or bleeding in the past year;
* subject has not had any hormonal agents or devices within 4 weeks prior to enrollment (Mirena is acceptable. n.b. Mirena can cause irregular menstrual cycles; however, this would not be exclusionary for the purposes of this protocol);
* subject, if a woman of child-bearing potential, must have had two consecutive normal menstrual cycles immediately prior to enrollment;
* subject must be in good health as determined by a physician (i.e., via medical history at the Pretreatment Screening Period, physical examination and screening laboratory results at the Pretreatment Screening and Baseline Periods);
* subject must weigh at least 50 kg and have a Body Mass Index (BMI) between 18 and 30, inclusive, at Pretreatment Screening Period;
* subject must have had normal clinical laboratory test results or, if abnormal, the clinical laboratory tests are not clinically significant in the Investigator's opinion, during the Pretreatment Periods;
* subject must have negative drug and alcohol toxicology screens during the Pretreatment Screening Period; and
* subject must have negative HIV antibody and hepatitis panel screening results during the Pretreatment Screening Period.
* For men over 44 years of age, Prostate Specific Antigen (PSA) is less than or equal to 2.0 ng/mL;
* For women over 44 years of age, mammography (within 3 months prior to Day 1) and pelvic ultrasound, with results showing no significant abnormality in the opinion of the Investigator, and specifically no suggestion of breast or endometrial neoplasm;
* subject must have Protein C and Protein S activity levels above the lower limit of normal;
* subject must have a negative test for Factor V Leiden.

Exclusion Criteria:

* subject has a history of any chronic condition of clinical significance, in the Investigator's opinion, that would preclude participation in the study (e.g. any clinically significant cardiovascular, hepatic, renal, or gastrointestinal abnormality);
* subject has a total bilirubin level greater than 0.9 mg/dL, a conjugated bilirubin greater than 0.4 mg/dL or an unconjugated bilirubin greater than 0.8 mg/dL at Screening; Fasting cholesterol level at screening is greater than 280 mg/dL; Fasting triglyceride level at screening is greater than 1.5 x the upper limit of normal;
* subject has any history of thromboembolic events or estrogen-dependent benign or malignant neoplasm;
* subject has resting systolic blood pressure >140 mm Hg or <90 mm Hg, or diastolic blood pressure >90 mm Hg or <60 mm Hg during the Pretreatment Screening Period;
* subject has a resting pulse >100 beats/minute or <45 beats/minute during the Pretreatment Screening Period;
* subject does not have a normal 12-lead electrocardiogram (ECG) during the Pretreatment Screening Period, or, if abnormal, the ECG is clinically significant in the opinion of the Investigator;
* subject is unwilling to comply with study rules, including attempting to void at specified times (prior to ECG time points) or maintain quiet, undistracted, awake, motionless supine posture during specified time points or exhibits anxious, excitable, hostile, or emotionally reactive affect;
* subject cannot tolerate a controlled, quiet study conduct environment, including avoidance during specified time points of music, TV, movies, games and activities that may cause excitement, emotional tension or arousal;
* subject has a history of sudden cardiac death in the immediate family, or a personal history of cardiac disease, treated hypertension, congestive heart failure, or unexplained syncope;
* subject has a previous history of cancer, other than basal cell carcinoma or stage 1 squamous cell carcinoma that has not been successfully treated;
* subject has taken any prescription or over-the-counter medication within 1 week prior to the Pretreatment Baseline Period (Day -1), or anticipates the need for any medication during the course of the study;
* subject has a history of intolerance to estrogen medication;
* subject has a history of substance abuse, drug addiction, or alcoholism within 3 years prior to the Pretreatment Baseline Period. (According to the DSM IV, alcohol abuse is defined as average consumption of more than 4 alcoholic drinks per day.);
* subject anticipates an inability to abstain from alcohol, caffeine or Yerba mate tea, or from grapefruit, grapefruit juice, or flavonoid-rich foods from 48 hours prior to the administration of study medication and throughout the duration of the study. Coca tea and mate de coca are not allowed within 1 week prior to Screening;
* subject has a history of smoking or any use of a tobacco product within 6 months prior to the Pretreatment Baseline Period;
* subject has donated blood or blood products within 30 days prior to the Pretreatment Baseline Period;
* subject is mentally unstable or is incapable of being compliant with the protocol;
* subject has received an investigational test substance within 60 days prior to the administration of investigational test article, or anticipates receiving any investigational test substance other than S-equol during the course of this study; or
* subject has been previously enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 14 days

SECONDARY OUTCOMES:
Total and free S-equol concentrations | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bianchi, MD, Principal Investigator — Syneos Health
Locations (1):
- Charles River, Tacoma, Washington, United States